CLINICAL TRIAL: NCT01550913
Title: Sober Network IPT for Perinatal Women With Comorbid Substance Use and Depression
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Caron Zlotnick, Director of Behavioral Medicine Research, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34DA030428-01A1 (NIH); R34DA030428-01A1 (NIH)
Record Dates: First submitted 2012-03-05; First posted 2012-03-12 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Perinatal Depression, Substance Use
Keywords: Substance use; perinatal depression; pregnant
MeSH Terms: conditions — Substance-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sober Network IPT (Experimental): Participants are assigned to Sober Network Interpersonal Psychotherapy (IPT)
  Interventions: Behavioral: Sober Network Interpersonal Psychotherapy (IPT)
- Treatment as Usual (Other): Participants are assigned to have Treatment as Usual
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Sober Network Interpersonal Psychotherapy (IPT) — IPT will be administered in 16 group 90-minute sessions over 18-20 weeks and 3 individual sessions (at the beginning, middle and end of treatment). These sessions will focus on improving your relationships with others, building sober relationships, setting goals, and increasing coping skills.
  Arms: Sober Network IPT
Other: Treatment as Usual — Women in the treatment as usual condition will either be referred to appropriate treatment in the community or continue their current substance use treatment.
  Arms: Treatment as Usual

SUMMARY:
This study will evaluate the effectiveness of Sober Network Interpersonal Psychotherapy (IPT) in treating women with depression and comorbid substance abuse.

DETAILED DESCRIPTION:
Substance use disorder (SUD) and major depressive disorder (MDD) are significant and interconnected public health problems facing women, especially perinatal women. Perinatal women with co-occurring SUD-MDD are of public health concern because they face numerous neonatal and obstetrical risks in addition to the emotional distress, impairment, and adverse health effects associated with these disorders. MDD is common in women with SUD, often does not remit with SUD treatment, increases the risk of poor SUD treatment outcome, and should be treated. Despite the serious morbidity associated with both SUD and MDD in perinatal women and despite the consensus among perinatal researchers that there is a need for population-specific treatments that address the unique set of challenges associated with this period of a women's life, virtually no interventions have been developed or tested to address the specific needs of perinatal women with comorbid substance use and depression. Furthermore, many tests of existing treatments for SUD-MDD in any population have demonstrated limited efficacy for at least one of the two disorders.

The investigators propose to pilot test a novel 18-20 week group treatment for SUD-MDD, Sober Network Interpersonal Psychotherapy(IPT), which focuses on network support strategies for SUD (i.e., enhancement of active sober support) within a broader Interpersonal Psychotherapy (IPT) framework. IPT is the treatment of choice for MDD in perinatal populations. Sober network support is theoretically consistent with IPT and has been identified as an empirically supported mechanism of change of many efficacious SUD treatments. Interpersonal difficulties not only affect MDD, but are also strong predictors of SUD relapse in women. A social/interpersonal approach to SUD-MDD may be highly efficacious for and relevant to the needs of perinatal women because specific interpersonal challenges become more salient during the perinatal period. Pilot work (supported by Dr. Johnson's NIDA K23), has shown an IPT-based treatment to be feasible, acceptable, and efficacious for MDD among women prisoners with SUD-MDD, another vulnerable population with multiple needs. Thus, Sober Network IPT integrates a validated treatment for perinatal MDD with empirically supported SUD principles, using proposed mechanisms that are particularly relevant to the perinatal period and to our target population.

The purposes of this R34 Exploratory Research proposal are to (a) integrate network support strategies for SUD into an IPT framework to create Sober Network IPT for perinatal women with substance use and MDD (b) to collect preliminary data on its feasibility, acceptability, and initial efficacy within a clinical setting in collaboration with community therapists. Attempting to obtain a definitive effect size estimate is not an intended outcome of an R34 given the limited sample sizes typically supportable under this mechanism. The investigators will, however, collect preliminary information to explore potential treatment differences and likely effect size ranges. Findings from this proposal will lay the groundwork for a larger clinical trial.

The development aims of this R34 proposal are to:

1. Adapt IPT to Sober Network IPT for perinatal women with substance use and MDD.
2. Develop, implement, and evaluate a therapist training program and competence and adherence scales.
3. Improve the clarity, content, acceptability, and feasibility of Sober Network IPT using information gathered from two focus groups and a small open trial (n = 6) of perinatal women with substance use and MDD.

The pilot study aims of this R34 proposal are to:

1. Conduct a randomized pilot trial in a sample of 50 women who meet criteria for substance use and MDD during pregnancy or within one year postpartum to demonstrate the feasibility and acceptability of the proposed recruitment methods and research design, of the therapist training methods, and of delivering the Sober Network IPT treatment.
2. Examine preliminary evidence for the hypotheses that, relative to treatment-as-usual, Sober Network IPT will result in:

   * Fewer heavy drinking/drug using days through the 3 month follow-up (primary).
   * Reduced depressive symptoms at post-treatment and 3 month follow-up (primary).
   * Improved sober support and social support (secondary).
3. Explore the feasibility of using fetal, neonatal and infant outcomes and engagement in health prevention activities (such as immunization and well-child visits) as secondary outcomes in a subsequent trial.

As a result of this R34 Exploratory Research Project, the investigators will have adapted IPT into Sober Network IPT, a novel treatment approach for perinatal women with substance use and MDD, tested its feasibility, acceptability, and initial efficacy with an eye toward dissemination (see D2.13), and the investigators will be prepared to test its efficacy in future R01 clinical trials. From a longer term perspective, this program of research will advance clinical care and research endeavors for perinatal women with substance use and MDD; underserved women with clinical concerns that are of great public health significance. Furthermore, if Sober Network IPT is found to be efficacious in our vulnerable target population, the investigators anticipate that it could hold promise for a more heterogeneous substance use and MDD population.

ELIGIBILITY:
Inclusion Criteria:

1. pregnant or has delivered in the past year
2. reports the use of an illegal drug and/or consumption of 4 or more drinks on one occasion within the last 6 months; if postpartum, report the use of an illegal drug and/or consumption of 4 or more drinks on one occasion or 7 or more drinks in a week within the last 6 months; if pregnant, report the use of an illegal drug within the last 6 months and/or the consumption of 2 or more drinks in one month while pregnant, along with a history of consumption of 4 or more drinks on one occasion or 7 or more drinks in a week within 3 months pre-pregnancy
3. meets DSM-IV criteria of current Major Depressive Disorder (MDD) by Structured Clinical Interview for the DSM-IV(SCID) interview;
4. has a 17-item Hamilton Rating Scale for Depression (HRSD) score > 16, indicating moderate to severe depression;
5. is between 18 and 50 years old; and
6. is able to speak and read English sufficiently to be able to complete the study procedures

Exclusion Criteria:

1. meets lifetime criteria for:

   * bipolar disorder
   * a primary psychotic disorder
   * anorexia nervosa
   * bulimia nervosa
2. has started an SUD or MDD medication dose within the 8 weeks prior to enrollment
3. is imminently suicidal

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2011-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in heavy drinking/drug using days at 3 months | up to 3 months post-treatment
  Using the Timeline Followback, participants will report their daily use in the time period between each interview (intake, 6 weeks, 12 weeks, 18-20 weeks and 3 months post treatment). The number of heavy drinking/drug using days reported at intake will be compared to the number reported at the followup assessments.
Change from baseline in depressive symptoms at 18-20 weeks | baseline and 18-20 weeks
  The total score of the Hamilton Rating Scale for Depression from intake will be compared to the total score at the 18-20 week assessment to show a reduction in the depressive symptoms.
Change from baseline in depressive symptoms at 3 months | baseline and 3 months post-treatment
  The total score of the Hamilton Rating Scale for Depression from intake will be compared to the total score at the 3 month followup assessment to show a reduction in the depressive symptoms.

SECONDARY OUTCOMES:
Change from baseline in Sober and social support at 3 months | up to 3 months post-treatment
  Using the total score of the Multidimensional Scale of Perceived Social Support (MSPSS) reported at the intake and at the 3 month followup the improvement in social and sober support will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Caron Zlotnick, PhD, Principal Investigator — Women and Infants Hospital of Rhode Island
Locations (1):
- Women and Infants Hospital of Rhode Island, Providence, Rhode Island, United States